CLINICAL TRIAL: NCT03294577
Title: A Phase 3, Randomized Study to Evaluate Plinabulin Versus Pegfilgrastim in the Prevention of Severe Neutropenia in Breast Cancer Patients Receiving Myelosuppressive Chemotherapy With Docetaxel, Doxorubicin, and Cyclophosphamide (TAC) (Protective 2)
Brief Title: Plinabulin vs. Pegfilgrastim in Prevention of TAC Induced Neutropenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BeyondSpring Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BPI-2358-106 phase 3
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Plinabulin; Pegfilgrastim; Chemotherapy induced neutropenia; bone pain
MeSH Terms: interventions — pegfilgrastim; Granulocyte Colony-Stimulating Factor; NPI 2358; Docetaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Plinabulin is masked using a double-dummy design. Docetaxel/Doxorubicin/Cyclophasphamide administration is not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAC + Pegfilgrastim (Active Comparator): Phase 3:TAC + Pegfilgrastim (6 mg)+ D5W placebo
  D5W Placebo: 250 ml D5W to match the administration of plinabulin diluted in 250 ml D5W
  Interventions: Drug: Pegfilgrastim; Other: D5W Placebo; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)
- TAC + Pegfilgrastim + Plinabulin (Experimental): Phase 3: TAC+ Plinabulin (40 mg) + Pegfilgrastim (6 mg)
  Interventions: Drug: Plinabulin; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)

INTERVENTIONS:
Drug: Pegfilgrastim — PEGFILGRASTIM is a long-acting granulocyte colony-stimulating factor that stimulates the growth of neutrophils, to reduce the incidence of fever and infection in patients with certain types of cancer who are receiving chemotherapy that affects the bone marrow.
  Other Names: Neulasta; G-CSF
  Arms: TAC + Pegfilgrastim
Drug: Plinabulin — Plinabulin (BPI-2358) is a synthetic, low molecular weight, new chemical entity that belongs to the diketopiperazine class of compounds. Plinabulin is intended for intravenous (IV) infusion and is diluted in D5W and administered for 30 minutes (± 5 minutes).
  Other Names: BPI-2358; NPI-2358
  Arms: TAC + Pegfilgrastim + Plinabulin
Other: D5W Placebo — Placebo 250 ml D5W to match the administration of plinabulin diluted in 250 ml D5W
  Arms: TAC + Pegfilgrastim
Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC) — Docetaxel is a type of chemotherapy medicine called an taxane. Doxorubicin is a type of chemotherapy medicine called an anthracycline. Cyclophosphamide is a type of chemotherapy medicine called an alkylating agent.
  Other Names: Taxotere; Adriamycin; Cytoxan

SUMMARY:
The primary purpose of this study is to compare the percentage of patients with Duration of Severe Neutropenia (DSN) =0 in patients treated with:

Docetaxel, doxorubicin, and cyclophosphamide (TAC) + pegfilgrastim versus Docetaxel, doxorubicin, and cyclophosphamide (TAC) + combination plinabulin/pegfilgrastim

Severe neutropenia is an absolute neutrophil count (ANC) <0.5 × 10^9/L.

Docetaxel, doxorubicin, and cyclophosphamide (TAC) will be used as the chemotherapy in this study.

DETAILED DESCRIPTION:
This is a multi-center randomized study, double-blind phase 3 trial. Approximately 222 patients are planned to be enrolled in Phase 3.

Docetaxel, doxorubicin, and cyclophosphamide (TAC) will be used as the chemotherapy in this study. These agents are among the most active and commonly used chemotherapeutic agents employed for treating patients with breast carcinoma. In particular, TAC chemotherapy has been used for the adjuvant treatment of HER2 negative early breast cancer patients with node positive disease as well as for node negative breast cancer patients who have a high risk of recurrence.

Plinabulin is a novel small molecule that is being developed for the mitigation of chemotherapy-induced neutropenia. Administered by IV infusion on the same day of (approximately 1 hour after) chemotherapy (TAC), plinabulin will be given in a single dose per cycle. Plinabulin is being studied to see if it is a convenient alternative to G-CSF, pegfilgrastim, for the prevention of chemotherapy-induced neutropenia.

In this trial, treatment will be double blinded, approximately 222 patients with breast cancer are expected to be enrolled. Patients are randomly assigned to one of the treatment arms, with 111 patients enrolled in each arm, with the arm designation and planned intervention as follows:

Arm 1: TAC + pegfilgrastim (6.0 mg) + placebo matching plinabulin.

Arm 2: TAC + pegfilgrastim (6.0 mg) + plinabulin (40 mg).

Cycles 1 to 4 will consist of TAC (or TC for Cycles 2 to 4) administered IV on Day 1 every 21 days. Patients will receive a single dose of plinabulin or placebo IV over 30 minutes (±5 minutes) in a double blinded manner, 30 minutes after the end of the TAC (or TC for Cycles 2 to 4) infusion. On Day 2 of each cycle (≥24 hours after completing chemotherapy), all patients will receive a single dose of pegfilgrastim (6.0 mg).

The long-term safety follow-up through patients contacts by phone calls, letters or electronic means; or medical records reviews will be conducted to all subjects approximately every 6 months up to 5 years to monitor long term safety of plinabulin.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are at least 18 years of age at the time of signing the informed consent form.
2. In the opinion of their treating oncology investigator, are candidates for at least 4 cycles of chemotherapy with TAC (docetaxel, doxorubicin, & cyclophosphamide).
3. Patients who are candidates for adjuvant or neoadjuvant TAC will meet all of the following criteria:

   * Biopsy-proven, early stage (Stage I and II) and Stage III breast cancer, and
   * Have had no prior chemotherapy.
4. Pathological confirmation of cancer is required.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Have life expectancy of 3 months or more.
7. Laboratory results provided by the central laboratory within 14 days prior to study drug administration within noted ranges, per study protocol (local laboratories may be accepted on a case by case basis after discussion with the medical monitor; however in this case central laboratories must also be taken within the screening time window)
8. Prothrombin time (PT) and International Normalized Ratio (INR) ≤1.5 × ULN, activated partial thromboplastin time (PTT) ≤1.5 × ULN, based on central laboratory results.
9. Women of childbearing potential have a negative pregnancy test at screening.

Exclusion Criteria:

1. History of myelogenous leukemia, myelodysplastic syndrome, or sickle cell disease.
2. Use of strong CYP3A4, CYP2D6 or P-glycoprotein (P-gp) inhibitors and inducers, within 14 days of the first administration of study drug and for the duration of the study.
3. Received an investigational agent or tumor vaccine within 2 weeks before the first dose of study drug; patients must have recovered from toxicity of prior treatment and have no >Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) treatment emergent adverse events (TEAE).
4. Receiving any concurrent anticancer therapies (including concomitant anti-HER2/neu agents such as trastuzumab [Herceptin®], trastuzumab emtansine [TDM 1, Kadcyla®], pertuzumab [Perjeta®], lapatinib [Tykerb®]).
5. Received a prior bone marrow or stem cell transplant.
6. Have a co-existing active infection or received systemic anti-infective treatment within 72 hours before the first dose of study drug.
7. Concurrent or prior radiation therapy within 4 weeks before the first dose of study drug.
8. Chronic use of filgrastim, pegfilgrastim, or any bioequivalent (biosimilar) for severe chronic neutropenia or other chronic neutropenia syndrome.
9. Presence of any serious or uncontrolled illness including, but not limited to: uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled arterial thrombosis, symptomatic pulmonary embolism, and psychiatric illness that would limit compliance with study requirements or any other conditions that would preclude the patient from study treatment as per the discretion of the Investigator.
10. Significant cardiovascular history:

    * Cardiac ventricular dysfunction inhibiting the patient's ability to receive 4 cycles of doxorubicin.
    * History of myocardial infarction or ischemic heart disease within 1 year (within a window of up to 18 days less than 1 year) before first study drug administration
    * Uncontrolled arrhythmia
    * History of congenital QT prolongation
    * Electrocardiogram (ECG) findings consistent with active ischemic heart disease
    * New York Heart Association Class III or IV cardiac disease;
    * Uncontrolled hypertension: blood pressure consistently >150 mm Hg systolic and > 100 mm Hg diastolic in spite of antihypertensive medication
11. History of hemorrhagic diarrhea, inflammatory bowel disease, or active uncontrolled peptic ulcer disease. (Concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
12. Any other active malignancy requiring active therapy.
13. Known human immunodeficiency virus (HIV) seropositivity.
14. Active Hepatitis B virus (HBV) infection which requires antiviral treatment or the patient has detectable Hepatitis B surface Antigen (HBsAg); hepatitis B surface antibody (anti-HBs) without detectable HBsAg does not exclude patients from the study. Hepatitis C infection (Hepatitis C antibody reactive) which requires treatment also excludes patients from the study.
15. Female patient who is pregnant or lactating.
16. Use of prophylactic antibiotics.
17. Unwilling or unable to comply with procedures required in this protocol.
18. History of allergy to any of the study drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with Duration of Severe Neutropenia (DSN) =0 | Duration of Grade 4 neutropenia assessed during the first cycle (21 days)
  DSN is defined as Days of Grade 4 Neutropenia (ANC less than 0.5 X 109/L)

SECONDARY OUTCOMES:
Mean DSN assessment | From day 1 to day 8 in first cycle (21 days)
  DSN is defined as Days of Grade 4 Neutropenia (ANC less than 0.5 X 109/L)
Mean ANC nadir | Duration of first cycle (21 days)
  record and evaluate the lowest ANC value
Percentage of Patients without grade 3 and grade 4 neutropenia | Duration of first cycle (21 days)
  ANC less than 1 x 109/L and above 0.5x 109/L is defined as grade 3 neutropenia. ANC less than 0.5 X 109/L is defined as grade 4 neutropenia.
Mean DSN assessment within 15 days | From day 1 to day 15 in the first cycle (21 days)
  To evaluate the effect of Plinabulin related to DSN within 15 days
Average change in bone pain | From -1 day over the observational period
  Record the bone pain score from the numerical rating scale (NRS)
Rate of composite risks | Duration of all 4 cycle (21 days)
  Composite risks includes infection, FN, hospitalization, significant disability, life threatening and death
Percentage of patients with relative dose intensity < 85% | Duration of all 4 cycle (21 days)
  Assess the percentage of patients with RDI < 85%

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Blayney, M.D., Study Chair — Stanford University School of Medicine - Cancer Institute
Locations (20):
- China (7):
  - No. 1 Banshandong Road, Hangzhou, Gongshu District
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University Breast Oncology, Guangzhou, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin, Harbin
  - Fourth Hospital of Hebei Medical University Breast cancer department, Shijiazhuang, Hebei
  - China-Japan Union Hospital of Jilin University Tumor department of Hematology, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Shenyang
- Ukraine (13):
  - Dnipropetrovsk City Multifunctional Hospital #4 Oncology Department, Dnipro
  - Prykarpatskiy Regional Oncological Center, Ivano-Frankivsk
  - Regional Clinical Oncology Center, Kharkiv
  - V.T. Zaycev Institute, Kharkiv
  - Kirovograd Regional Oncological Center, Kropyvnytskyi
  - Public Institution Kryvyi Rih Oncology Center, Krutyi Bereh
  - Hemotherapy Department, Kyiv
  - Kyiv City Clinical Oncological Center, Kyiv
  - Lviv State Oncological Regional, Lviv
  - Odessa regional clinical hospital Thoracic Surgery Department Academician Zabolotnoho, Odesa
  - Zakarpattia Regional Clinical Oncology Center, Uzhhorod
  - Vinnytsya Regional Clinical Oncology Dispensary, Vinnytsia
  - Zaporizhia Regional Clinical Oncology Dispensary, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No